CLINICAL TRIAL: NCT02486848
Title: Minoxidil Dose Response Study in Females Identified Through IVD Testing as Non-Responders to 5% Topical Minoxidil
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Maja Kovacevic, MD (Industry)
Responsible Party: Sponsor-Investigator, Maja Kovacevic, MD, Clinical Researcher, Applied Biology, Inc.
Organization: Applied Biology, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FI-DRUG-MINOXIDIL-001
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Female Pattern Hair Loss; Androgenetic Alopecia
Keywords: Hairloss; Female Pattern Hair Loss; Androgenetic Alopecia; Minoxidil
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% Topical Minoxidil Solution (Placebo Comparator): 5% Topical Minoxidil Solution
  Interventions: Drug: 5% Topical Minoxidil Solution
- 15% Topical Minoxidil Solution (Active Comparator): 15% Topical Minoxidil Solution
  Interventions: Drug: 15% Topical Minoxidil Solution

INTERVENTIONS:
Drug: 5% Topical Minoxidil Solution — 5% Topical Minoxidil Solution
  Arms: 5% Topical Minoxidil Solution
Drug: 15% Topical Minoxidil Solution — 15% Topical Minoxidil Solution
  Arms: 15% Topical Minoxidil Solution

SUMMARY:
5% topical minoxidil is the maximum dosage approved by the US FDA for the treatment of female pattern hair loss. While topical minoxidil exhibits a good safety profile, the efficacy in the overall population is relatively low i.e., 30-40% re-grow hair.

The primary purpose of this study is to assess if a higher dosage of topical minoxidil dosage (15%) will increase the number of responders among female subjects that have been identified through IVD testing as non-responders to 5% topical minoxidil.

DETAILED DESCRIPTION:
Approximately, 40% of women suffer from female pattern hair loss by the age of 55. Currently, there is only one drug approved by the US FDA for the treatment of female pattern hair loss (AGA) - topical minoxidil.

5% topical minoxidil is the maximum dosage approved by the US FDA for the treatment of female AGA. While topical minoxidil exhibits a good safety profile, the efficacy in the overall population is relatively low i.e., 30-40% re-grow hair.

Minoxidil is a pro-drug. To elicit a clinical response, minoxidil must be converted to its active form minoxidil sulfate by a sulfotransferase enzyme found in hair follicles. The investigators have developed an in-vitro diagnostic test that correctly identifies, prior to initiating therapy, 95.9% of non-responders to 5% topical minoxidil. The diagnostic test analyzes the sulfotransferase enzymatic activity in hair follicles to determine if a sufficient amount of minoxidil will be converted to the active form required to induce hair growth. Subjects with low enzymatic activity experience little or no therapeutic benefit and a reduced frequency of adverse events.

Consequently, the investigators hypothesize that in subjects with low enzymatic activity (i.e., low minoxidil metabolizers) an increased minoxidil dosage will elicit a therapeutic response with little or no increase in the frequency of adverse events. It is thus the primary purpose of this study to assess if a higher dosage of topical minoxidil dosage (15%) will increase the number of responders among female subjects that have been identified through IVD testing as non-responders to 5% topical minoxidil.

ELIGIBILITY:
Inclusion Criteria:

* Females in overall good health
* Age: 18 to 55
* Female pattern hair loss (Sinclair 2-4)
* Willing to have a mini dot tattoo placed in the target area of the scalp
* Willing to maintain the same hair style, color, shampoo and hair products use, and approximate hair length throughout the study
* Able to give informed consent
* Non-responder to 5% minoxidil as determined by the MX-IVD test i.e., low minoxidil metabolizer
* Able to comply with the study requirements for 24 consecutive weeks
* Willing to use an adequate method of birth control (if applicable)
* Negative urine pregnancy test

Exclusion Criteria:

* Previous adverse event from topical minoxidil treatment
* History of hypotension
* Uncontrolled hypertension
* Use of any hypertensive drugs
* Pregnant, nursing, or planning a pregnancy during the study
* Prior hair transplant
* Uses wigs or hair weaves
* Have used minoxidil (topical or oral) anytime during the past 6 months
* Chronic scalp disorders that require medications
* Uses medication known to cause hair thinning such as Coumadin and anti-depressants/anti-psychotics
* Folliculitis
* Scalp psoriasis
* Seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopilaris
* Enrolled in any other medical study or has been enrolled in any medical study in the past 30 days
* Responder to 5% minoxidil as determined by the MX-IVD test

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Target Area Hair Count | baseline to week 24
  Target Area Hair Count. Number of hairs measured in the target area by macrophotography
Subjects Ratings | baseline to week 24
  Subjects Ratings

SECONDARY OUTCOMES:
Target Area Hair Count | baseline to week 12
  Target Area Hair Count. Number of hairs measured in the target area by macrophotography.
Expert Panel Global Photography Assessment | baseline to week 24
  Treatment efficacy evaluated by expert panel review of global photographs assessing hair regrowth

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kovacevic, MD, Principal Investigator — University of Rome, Italy ("G. Marconi")
Locations (1):
- Istituto Scienze Dermatologiche, Florence, Tuscany, Italy

REFERENCES:
- [Background] Roberts J, Desai N, McCoy J, Goren A. Sulfotransferase activity in plucked hair follicles predicts response to topical minoxidil in the treatment of female androgenetic alopecia. Dermatol Ther. 2014 Jul-Aug;27(4):252-4. doi: 10.1111/dth.12130. Epub 2014 Apr 28. PMID 24773771
- [Background] Goren A, Castano JA, McCoy J, Bermudez F, Lotti T. Novel enzymatic assay predicts minoxidil response in the treatment of androgenetic alopecia. Dermatol Ther. 2014 May-Jun;27(3):171-3. doi: 10.1111/dth.12111. Epub 2013 Nov 27. PMID 24283387
- [Background] Buhl AE, Waldon DJ, Baker CA, Johnson GA. Minoxidil sulfate is the active metabolite that stimulates hair follicles. J Invest Dermatol. 1990 Nov;95(5):553-7. doi: 10.1111/1523-1747.ep12504905. PMID 2230218
- [Background] Messenger AG, Rundegren J. Minoxidil: mechanisms of action on hair growth. Br J Dermatol. 2004 Feb;150(2):186-94. doi: 10.1111/j.1365-2133.2004.05785.x. PMID 14996087